CLINICAL TRIAL: NCT02981901
Title: Optimisation of Disease Management in Patients With Epithelial Ovarian Cancer in France
Acronym: Ovaire01
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Collaborators: Cancer Côte d'or registry (Unknown); Cancer Calvados registry (Unknown)
Responsible Party: Sponsor
Other Study IDs: Ovaire01
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with ovarian epithelial cancer: Ovarian epithelial cancer diagnosed in 2012
  Interventions: Other: Patient with ovarian epithelial cancer

INTERVENTIONS:
Other: Patient with ovarian epithelial cancer

SUMMARY:
No structured organization for ovarian first line management emerges in France. Management across France seems to depend on regional contexts.

Regions display no specific organization or delineate regional network for the ovarian cancer management or report centralized management revolving around referent centers. These different templates present a major problem in identifying differences, costs and benefit.

To deal with this issue the Investigators propose a health economic evaluation based on cost-effectiveness analyses, completed with a budget impact analysis. This study will investigate the cost-effective management of patients with initial ovarian cancer using databases representative of different parts of French territories.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian epithelial cancer initially diagnosed in 2012
* Age > 18 years old
* Residency in France (Rhône-Alpes region, District of Calvados and Cotes d'Or)
* First-line ovarian epithelial cancer

Exclusion Criteria:

* Relapsed ovarian epithelial cancer
* Non epithelial ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with ovarian epithelial cancer diagnosed in 2012
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incremental cost-effectiveness ratio expressed in cost per relapse-free year gained | 2 years after diagnosis
  To perform a cost-effectiveness analysis in order to evaluate the most efficient organization for ovarian cancer in 1st line ot treatment

SECONDARY OUTCOMES:
Incremental cost-effectiveness ratio expressed in cost per QALY(Quality-Adjusted Life Year) gained. | 2 years after diagnosis
Budget impact analysis | 2 years after diagnosis
  Cost assessment performed retrospectively for each patient: hospital stays, visits and other health-related costs will be identified and measured based on the French national Health Insurance perspective.
  QALY (Quality-Adjusted Life Year)
Relapse-free survival (RFS) | RFS will be assessed 2 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle RAY-COQUARD, PU-PH, Principal Investigator — Centre Leon Berard
Locations (3):
- France (3):
  - Calvados registry, Caen
  - Côte d'or registry, Dijon
  - Oveval, Lyon